CLINICAL TRIAL: NCT03244748
Title: Effect of Amiodarone After Ischemic Ventricular Tachycardia Ablation
Brief Title: Amiodarone Usage After Ischemic Ventricular Tachycardia Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Principal Investigator, Fırat Özcan, Associate Professor, Yuksek Ihtisas Hospital
Other Study IDs: ozcan01
Record Dates: First submitted 2017-08-05; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Ischemic Cardiomyopathy; Ventricular Tachycardia; ICD Shock
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients underwent ablation and continued having amiodarone after the procedure
  Interventions: Procedure: Ventricular tachycardia ablation
- Group 2: Patients underwent ablation and not having amiodarone after the procedure
  Interventions: Procedure: Ventricular tachycardia ablation

INTERVENTIONS:
Procedure: Ventricular tachycardia ablation — Electrophysiologic procedure aims to ablate and terminate arrhythmia percutaneously

SUMMARY:
Ventricular Tachycardia ablation in ischemic cardiomyopathy patients is required procedure in cases when anti-arrhythmic drugs failed. The concern is if adjunctive continuation amiodarone after ablation is needed.

DETAILED DESCRIPTION:
Ischemic cardiomyopathy patients have implantable cardioverter defibrillators (ICD) to prevent arrhythmic deaths. Ventricular tachycardia (VT) events with frequent ICD interventions in ischemic cardiomyopathy patients is encountered frequently. Frequents ICD interventions is associated with worse outcomes. Anti-arrhythmic drugs ,mostly amiodarone, are given prevent ventricular arrhythmias and ICD interventions that may not be curative. Ablation of ventricular tachycardia is the suggested treatment when anti-drugs are without effect. After ablation of ventricular arrhythmia the continuation of amiodarone is not well elucidated.

In this study we aimed to enroll ischemic cardiomyopathy patients having frequent ICD interventions despite medical treatment. VT ablation is performed and patients divided into two groups; group one continues having amiodarone after ablation, group two does not have amiodarone after ablation. Both groups will be compared in terms of recurrence and death.

ELIGIBILITY:
Inclusion Criteria:

Ischemic cardiomyopathy patients applied with frequent ICD interventionor electrical storms and having ejection fraction below 50%. Frequent ICD defined as more than 1 ICD intervention within month. Electrical storm defined as more than 2 ICD intervention within one day.

Exclusion Criteria:

Patients with cardiomyopathies other than ischemic etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enroll ischemic heart failure patients who had frequent ventricular arrhythymias causing multiple shocks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | six months
  Death, ICD intervetion

CONTACTS AND LOCATIONS:
Overall Officials: Firat Ozcan, MD, Principal Investigator — MD
Locations (1):
- Turkiye Yuksek Ihtisas Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No